CLINICAL TRIAL: NCT05217875
Title: Prognostic of Dysfunctional Breathing in Long Covid: a Follow up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital du Valais (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01698
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Dysfunctional Breathing
Keywords: COVID-19; Dysfunctional breathing; Hyperventilation syndrome; Sighs; erratic breathing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dysfunctional breathing might participate to dyspnoea in long COVID-19. This study investigate the prognosis of patients diagnosed with dysfunctional breathing after SARS-CoV-2 infection in our center.

DETAILED DESCRIPTION:
Dysfunctional breathing (DB) with or without hyperventilation syndrome (HVS) as diagnosed using cardiopulmonary exercise test (CPET) was recently demonstrated as an important physiopathological mechanism of persistent dyspnoea in long COVID patients [1]. DB is characterized by specific ventilation pattern on CPET accompanied by respiratory discomfort and/or dyspnea at exercise [2]. Most patients with DB will have undergone some sort a specific physiotherapy retraining [3]. However the prognostic and the predictors of persistence/resolution of DB after severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection are unknown.

The aim of the study is to determine the prognostic of patients diagnosed with DB after SARS-CoV-2 infection, as well as prognosis factors and predictors of persistence/resolution of DB during a prospective follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* patients 14 years or more
* diagnosis of DB after SARS-CoV-2 at our long covid clinic using a combined approach of symptoms and CPET analysis in the hospitals of Sion, Martigny or Rennaz
* Inclusion between November 2020 and until the end of October 2021

Exclusion Criteria:

* Refusal to participate
* comorbidities preventing the CPET or PFT to be carried out

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients of 14 years or more diagnosed with DB after COVID-19 using a combined approach of symptoms and CPET in the Hospitals of Sion, of Martigny or Rennaz
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Persistence/resolution of dysfunctional breathing at follow-up visit | 6 to 9 monts from diagnosis
  defined by persistence/resolution of dyspnea, as compared with patient's baseline (equivalent level of dyspnea as before COVID-19).

SECONDARY OUTCOMES:
Change in ventilatory patterns (tidal volume [VT], breathing frequency [BF] at isowork as compared with baseline | 6 to 9 monts from diagnosis
Dispersion of VT and BF during the CPET | 6 to 9 monts from diagnosis
Change in ETCO2 and PaCO2 | 6 to 9 monts from diagnosis
Qualitative changes (increase/decrease/no change of DB pattern of CPET) | 6 to 9 monts from diagnosis
Score HADS changes | 6 to 9 monts from diagnosis
Score SF-36 changes | 6 to 9 monts from diagnosis
Specific symptom scale changes | 6 to 9 monts from diagnosis
Specific work capacity changes questions | 6 to 9 monts from diagnosis
Post-COVID Functional Status (PCFS) changes | 6 to 9 monts from diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier du valais romand, Martigny-Ville, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data upon reasonable requests